CLINICAL TRIAL: NCT02787772
Title: Abdominal Hernia in Cirrhotic Patients: Surgery or Conservative Treatment?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Wellington Andraus, Prof. PhD. MD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0937/09
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Liver Cirrhosis; Hernia; Ascites; Surgery
MeSH Terms: conditions — Liver Cirrhosis; Hernia; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elective Hernia Repair (Experimental): Elective abdominal wall hernia surgery was performed in randomized cirrhotic patients.
  Interventions: Procedure: Elective Hernia repair
- Clinical follow up (No Intervention): Cirrhotic patients were kept in clinical follow up concerning their abdominal wall hernia.
  If a complication occured at the hernia site (such as skin rupture, bowel strangulation,..) the patient underwent emergency hernia repair.

INTERVENTIONS:
Procedure: Elective Hernia repair — abdominal wall hernia repair using onlay mesh.
  Arms: Elective Hernia Repair

SUMMARY:
Cirrhotic patients have a high incidence of abdominal wall hernias. Ascites and sarcopenia are risk factors to development of bigger hernias and frequent need for urgent surgery due parietal complications. However, hernia surgery is usually delayed in cirrhotic patients because of high morbidity and mortality.

Methods: A prospective study of cirrhotic patients with abdominal wall hernia during January 2009 to November 2014. Demographics, characteristics of underlying liver disease, type of hernia, complications and mortality of 246 enrolled patients were collected. Elective hernia repair was performed in 57 unselected patients, 186 patients were kept in clinical follow up. During follow up urgent hernia surgery was performed when unavoidable

DETAILED DESCRIPTION:
Abdominal wall hernias are frequent in cirrhotic patients. The incidence of umbilical hernia´s reaches over 20% in compensated cirrhosis and even 40% in patients with ascites. Several risk factors explain the development of umbilical hernia in these patients, such as, increased intra-abdominal pressure caused by ascites; abdominal aponeurosis weakness due sarcopenia ; and recanalization of the umbilical vein. These hernias develop great hernial sacs, especially when ascites is present. All these risk factors also explain their high complication rate due to the development of pressure ulcers, skin rupture, ascites leak and bacterial peritonitis. Moreover pain is a common associated symptom.

Inguinal hernias also develop due to higher intra-abdominal pressure due to ascites; they often result in large hernia sacs reaching the scrotum. In addition such large hernias are responsible for reduced mobility and quality of life.

The ideal treatment would be to correct both the abdominal wall hernia and the underlying liver disease. However, there are insufficient liver´s donors, so the liver transplantation (LT) waiting list continuously grows. This explains why the majority of abdominal wall hernias in cirrhotic patients remain untreated for several years.

Therefore, most cirrhotic hernia patients are followed conservatively, the surgical treatment being reserved when complications occur. Such expectative attitude is explained by the high postoperative morbidity and mortality. Although, urgent surgery in such patients impose a higher morbidity and mortality compared to elective hernia surgery.

No prospective study is reported comparing the incidence of complications in cirrhotic hernia patients which are just observed or submitted to elective surgery. The aim of this study is to analyze the results of the surgical treatment of abdominal wall hernias in cirrhotic patients.

A prospective study was conducted in patients having documented cirrhosis and abdominal hernia that were followed at the Department of Liver Transplant of University of São Paulo during the period January 2009 to November 2014. All patients included in the study signed an informed consent. At that moment they were randomized for elective hernia repair or clinical follow-up accordingly to their Child-Pugh (CTP) status. Patients who developed local hernia complications during observation underwent emergency hernia surgery.

Cirrhosis was diagnosed by liver tests and confirmed with liver imaging or biopsy. Abdominal wall hernias were diagnosed by physical examination and ultrasound and/or CT scans when necessary.

All patients were managed for their liver disease using individualized laboratory tests, endoscopic and ultrasound work-up. Patients with decompensated liver disease were medically optimized using diuretics in order to control the ascites.

Variables studied were: age, sex, etiology of liver disease, CTP classification, MELD (model of end stage liver disease) score, ascites, need of paracentesis, diabetes mellitus, renal failure and abdominal hernia type, morbidity and mortality. In patients who underwent surgery length of hospital stay, post-operative complications, grade of complications accordingly Clavien and infection were also recorded. Post-operative mortality was considered up to 30-days. End points of the study were death, hernia recurrence or LT.

This study was approved by the Institutional Review Board of University of Sao Paulo.

Wait and see was the advocated policy before this study.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic liver disease (cirrhosis) and abdominal wall hernia.

Exclusion Criteria:

* patients who didn´t want to underwent hernia repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2009-01; Primary Completion 2014-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
mortality during follow up | 4 years
  Compare long-term survival in cirrhotic patients with abdominal wall hernia who underwent elective hernia repair or maintained in clinical follow up.

SECONDARY OUTCOMES:
post operative mortality | 30 days
  mortality after elective or urgent hernia repair in cirrhotic patients
post operative morbidity | 30 days
  post operative complications after elective or urgent hernia repair in cirrhotic patients
incidence of complications in patients clinical follow up | 4 years
  Incidence of hernia complications leading to emergency hernia repair

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belghiti J, Durand F. Abdominal wall hernias in the setting of cirrhosis. Semin Liver Dis. 1997;17(3):219-26. doi: 10.1055/s-2007-1007199. PMID 9308126
- [Background] Carbonell AM, Wolfe LG, DeMaria EJ. Poor outcomes in cirrhosis-associated hernia repair: a nationwide cohort study of 32,033 patients. Hernia. 2005 Dec;9(4):353-7. doi: 10.1007/s10029-005-0022-x. Epub 2005 Aug 27. PMID 16132187
- [Background] Marsman HA, Heisterkamp J, Halm JA, Tilanus HW, Metselaar HJ, Kazemier G. Management in patients with liver cirrhosis and an umbilical hernia. Surgery. 2007 Sep;142(3):372-5. doi: 10.1016/j.surg.2007.05.006. PMID 17723889
- [Background] Silva FD, Andraus W, Pinheiro RS, Arantes-Junior RM, Lemes MP, Ducatti Lde S, D'albuquerque LA. Abdominal and inguinal hernia in cirrhotic patients: what's the best approach? Arq Bras Cir Dig. 2012 Jan-Mar;25(1):52-5. doi: 10.1590/s0102-67202012000100012. English, Portuguese. PMID 22569980
- [Background] Mansour A, Watson W, Shayani V, Pickleman J. Abdominal operations in patients with cirrhosis: still a major surgical challenge. Surgery. 1997 Oct;122(4):730-5; discussion 735-6. doi: 10.1016/s0039-6060(97)90080-5. PMID 9347849
- [Background] Hassan AM, Salama AF, Hamdy H, Elsebae MM, Abdelaziz AM, Elzayat WA. Outcome of sublay mesh repair in non-complicated umbilical hernia with liver cirrhosis and ascites. Int J Surg. 2014;12(2):181-5. doi: 10.1016/j.ijsu.2013.12.009. Epub 2013 Dec 28. PMID 24378913
- [Background] Ammar SA. Management of complicated umbilical hernias in cirrhotic patients using permanent mesh: randomized clinical trial. Hernia. 2010 Feb;14(1):35-8. doi: 10.1007/s10029-009-0556-4. Epub 2009 Aug 29. PMID 19727551
- [Background] Andraus W, Pinheiro RS, Lai Q, Haddad LBP, Nacif LS, D'Albuquerque LAC, Lerut J. Abdominal wall hernia in cirrhotic patients: emergency surgery results in higher morbidity and mortality. BMC Surg. 2015 May 21;15:65. doi: 10.1186/s12893-015-0052-y. PMID 25990110
- [Background] de Goede B, Klitsie PJ, Lange JF, Metselaar HJ, Kazemier G. Morbidity and mortality related to non-hepatic surgery in patients with liver cirrhosis: a systematic review. Best Pract Res Clin Gastroenterol. 2012 Feb;26(1):47-59. doi: 10.1016/j.bpg.2012.01.010. PMID 22482525
- [Background] Oh HK, Kim H, Ryoo S, Choe EK, Park KJ. Inguinal hernia repair in patients with cirrhosis is not associated with increased risk of complications and recurrence. World J Surg. 2011 Jun;35(6):1229-33; discussion 1234. doi: 10.1007/s00268-011-1007-9. PMID 21365342